CLINICAL TRIAL: NCT06559228
Title: ConnectedNest: a Digital Platform Connecting Individuals With Cancer to Social Care
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024LS102
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ConnectedNest adults (Experimental): adults undergoing active cancer therapy or in cancer survivorship seen in multi-site oncology practices randomized to receive ConnectedNest
  Interventions: Other: ConnectedNest
- Standard of care adults (Active Comparator): adults undergoing active cancer therapy or in cancer survivorship seen in multi-site oncology practices randomized to receive standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: ConnectedNest — Participants will receive a secure message to register and download ConnectedNest's patient app, EmpowerNest. They will be asked to complete a set of modules at baseline through ConnectedNest to understand their health related social needs and programs available to meet those needs. They will receive basic training on the functionality and services available within the app and asked to use the app to identify and connect with needed social and community services for 90 days. Participants will be directed to complete a survey at baseline, 30, 60, and 90 days to collect patient-reported outcomes.
  Arms: ConnectedNest adults
Other: Standard of care — Participants will be directed to complete a survey at baseline, 30, 60 and 90 days to collect patient-reported demographics, cancer characteristics and outcomes metrics
  Arms: Standard of care adults

SUMMARY:
Social determinants of health (SDoH) such as housing instability, food insecurity, and financial burden largely shape the health and well-being of individuals, create health inequities, and drive a large portion of avoidable adverse health outcomes and healthcare costs. With new advancements in treatment and rising out-of-pocket expenses, individuals facing cancer are especially vulnerable to the adverse effects of SDoH. To address these barriers, a novel solution is needed to support oncology patients, clinical teams, and community-based organizations (CBOs) across the cancer continuum. In a Phase I contract award, XanthosHealth developed ConnectedNest, a novel electronic social care referral platform to screen for SDoH needs and connect individuals with cancer to social and community services provided by CBOs while engaging the oncology team in the SDoH referral process. Through additional funding, a pilot study was completed in Minneapolis, Minnesota, in partnership with Minnesota Cancer Alliance, involving the collaboration of 14 CBOs focused on cancer. 50 cancer survivors from these CBOs were enrolled to utilize the ConnectedNest platform for a 90-day duration. Our study involved the collection and analysis of crucial metrics related to patient and CBO engagement, SDoH needs, and the volume of feasible social care referrals. In Phase II, the technical features and integration capabilities of ConnectedNest will be enhanced based on learnings in Phase I and completed pilot study. The platform will be implemented and tested among patients seen at multiple oncology clinics, evaluating health outcomes of patients who use the platform.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 and over
* undergoing active cancer therapy or in survivorship
* must be able to read and write in English
* Seen in a participating Minnesota oncology clinic

Exclusion Criteria:

* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of self-reported social needs | Day 90
  change in the number of reported social needs from baseline (time of randomization) to day 90 after enrollment using the validated Accountable Health Communities Health-related social needs screening tool.
Reported social needs that are partially or completely met | Day 90
  change in the number of reported social needs that are partially or completely met from baseline (time of randomization) to day 90 after enrollment using the validated Accountable Health Communities Health-related social needs screening tool.

SECONDARY OUTCOMES:
Number of connections with needed social and community services with needed social and community services | Day 90
  Change in self-reported levels of distress using the National Comprehensive Cancer Network (NCCN) distress thermometer from baseline (time of randomization) to day 90 after enrollment
Quality of life | Day 90
  Change in self-reported quality of life from baseline (time of randomization) to day 90 after enrollment using the Functional Assessment of Cancer Survey-General
Satisfaction with Care | Day 90
  Change in self-reported satisfaction with care from baseline (time of randomization) to day 90 after enrollment using the Patient Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Helen Parsons, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States